CLINICAL TRIAL: NCT06215833
Title: Comparison of Emergence and Recovery Profile After Total Intravenous Anesthesia ( TIVA ) Vs Inhalational Anesthesia in Opioid Free Pediatric Tonsillectomy
Brief Title: Recovery of TIVA vs Inhalation in Pediatric Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Sayed, Principal Investigator, Assiut University
Other Study IDs: TIVA vs inhalation anesthesia
Record Dates: First submitted 2023-12-10; First posted 2024-01-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Best Technique for Pediatric Anesthesia
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group ( p ): This group will undergo anesthesia via total intravenous anesthesia using Propofol in induction and maintenance
  Interventions: Drug: Propofol
- Group ( s ): This group undergo anesthesia via total inhalational anesthesia using sevoflurane in induction and maintenance
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — All children will undergo anesthesia via Propofol bolus injection in induction then Propofol infusion in maintenance of anesthesia and will be given after total recovery, Cetal suppositories as postoperative analgesia
  Other Names: Cetal suppository
  Groups: Group ( p )
Drug: Sevoflurane — All children will undergo anesthesia via Sevoflurane will be given during induction then through maintenance of anesthesia and will be given after total recovery, Cetal suppositories as post operative analgesia
  Other Names: Cetal suppository
  Groups: Group ( s )

SUMMARY:
Compare recovery profile from TIVA and that of total inhalational anesthesia in ambulatory pediatric tonsillectomy and which strategy is more safe and less cost and more smooth in pediatric anesthesia.

DETAILED DESCRIPTION:
Complications in pediatric anesthesia can happen even in our modern hospitals with the most advanced equipment and skilled anesthesiologists.

Typical complications in pediatric anesthesia are respiratory problems , medication errors , difficulties with intravenous puncture , and pulmonal aspiration. In postoperative setting , nausea and vomiting , pain , emergence delirium can be mentioned as typical complications.

The choice of anesthetic agent and techniques can influence the occurrence of these complications and thus delay in discharge.

ELIGIBILITY:
Inclusion Criteria:

* child between 4 to 10 years
* without co morbidity
* ASA score 1
* mallampati score 1 and 2

Exclusion Criteria:

* child below 4 years and above 10 years
* child with co morbidity
* ASA score above 1
* mallampati score 3 and 4

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children planned for ambulatory tonsillectomy from primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
level of consciousness score | About 20 minutes after stopping anesthesia and emergence from anesthesia begin
  * Awake =2
  * Arousal with minimal stimulation =1
  * Responsive only to tactile stimulation =0
  * No score 0 is required & High score mean more safe and better method of anesthesia .
physical activity score | About 20 minutes after stopping anesthesia and emergence from anesthesia begin
  * Able to move on command =2
  * Some weakness in movement = 1
  * Unable to voluntarily move = 0
  * No score 0 is required & High score mean more safe and better method of anesthesia .
hemodynamic stability score | About 20 minutes after stopping anesthesia and emergence from anesthesia begin
  * Blood pressure < 15% of baseline MAP value =2
  * Blood pressure 15%-30% of baseline MAP value =1
  * Blood pressure < 30% below baseline MAP value =0
  * No score 0 is required & High score mean more safe and better method of anesthesia .
respiratory stability score | About 20 minutes after stopping anesthesia and emergence from anesthesia begin
  * Able to breathe deeply = 2
  * Tachypnea with good coughs =1
  * Dyspneic with weak cough = 0
  * No score 0 is required & High score mean more safe and better method of anesthesia .
Oxygen saturation score | About 20 minutes after stopping anesthesia and emergence from anesthesia begin
  * Maintain value > 90% on room air = 2
  * Requires supplemental O2 to maintain value > 90% = 1
  * So2 < 90% with supplemental O2 = 0
  * No score 0 is required & High score mean more safe and better method of anesthesia .
post operative pain score | About 20 minutes after stopping anesthesia and emergence from anesthesia begin
  * None or mild = 2
  * Moderate to severe pain controlled =1
  * Persistent severe pain = 0
  * No score 0 is required & High score mean more safe and better method of anesthesia .
post operative emetic score | About 20 minutes after stopping anesthesia and emergence from anesthesia begin
  * None or mild nausea with no active vomiting = 2
  * Transient vomiting =1
  * Persistent moderate to severe nausea and vomiting=0
  * No score 0 is required & High score mean more safe and better method of anesthesia .

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol